CLINICAL TRIAL: NCT00321854
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Clinical Trial to Examine the Efficacy and Safety of Early Pramipexole (PPX) Treatment Versus Delayed Pramipexole Treatment in Patients With New Onset Parkinson's Disease.
Brief Title: Study of (Mirapex) Pramipexole for the Early Treatment of Parkinsons Disease (PD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 248.595
Record Dates: First submitted 2006-05-03; First posted 2006-05-04 (Estimated); Results first posted 2010-01-26 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Early Pramipexole (Experimental): Patients were treated with pramipexole for 6 to 9 months then up-titrated to target dose of pramipexole (2.25 mg/day).
  Interventions: Drug: pramipexole
- Delayed Pramipexole (Experimental): Patients were treated with placebo for 6 to 9 months then up-titrated to target dose of pramipexole (2.25 mg/day).
  Interventions: Drug: pramipexole

INTERVENTIONS:
Drug: pramipexole

SUMMARY:
This is a double blind, placebo-controlled clinical trial of 15 months duration designed to examine early Mirapex (pramipexole) treatment vs. delayed Mirapex (pramipexole) treatment in patients with new onset Parkinsons disease

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent in accordance with Good Clinical Practice (GCP) and local legislation;
* Male or female patient with idiopathic Parkinson Disease (PD) confirmed by at least three of the following signs: resting tremor, bradykinesia, rigidity, and asymmetry (must have bradykinesia);
* Parkinsons disease newly diagnosed within the past 2 years;
* Patients with idiopathic PD characterized as Stage I-II by the Modified Hoehn and Yahr Scale who do not require PD medication and will not likely need PD medication for at least 6 months in the opinion of the investigator; Age 30 to 75 years at screening (Visit 1);
* Women of childbearing potential must have a negative serum Beta-HumanChorionGonadotropin (Beta-HCG) pregnancy test at the Screening (Baseline) visit unless surgically sterile or post-menopausal (last menstruation 12 months prior to signing Informed Consent). Women of childbearing potential must be using a medically accepted contraceptive method. Acceptable methods of birth control are limited to: Intra-Uterine Device (IUD), oral, implantable, or injectable contraceptives, estrogen patch, and double barrier method (spermicide + diaphragm); and Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Previous history of allergic response or complications with pramipexole (PPX) or its excipients;
* Atypical PD syndromes due to either drugs (e.g., metoclopramide, flunarizine) or metabolic disorders (e.g., Wilsons Disease), encephalitis, or degenerative diseases (e.g., progressive supranuclear palsy);
* The patient is currently on L-dopa, dopamine agonists or other PD medication at baseline;
* The patient has been on L-dopa, dopamine agonists or other PD medications for greater than 14 consecutive days prior to baseline;
* If on L-dopa, dopamine agonists or other PD medications prior to baseline, the patient stopped treatment less than 30 days prior to baseline;
* The patient has clinically significant abnormal laboratory values, and/or medical or psychiatric illness other than as seen in Parkinsons disease;
* The patient has a clinically significant deviation from normal in the physical examination other than as seen in Parkinsons disease;
* The patient has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery);
* History of stereotactic brain surgery;
* Surgery within 6 months of randomization, which in the opinion of the investigator, would negatively impact the patients participation in the study;
* History of active epilepsy (i.e., occurrence of a seizure) within the past year;
* Symptomatic orthostatic hypotension prior to randomization;
* Malignant melanoma or history of previously treated malignant melanoma;
* Patients who have received any of the following drugs (all time periods are calculated from randomization): Amantadine;
* Electroconvulsive therapy during 180 days preceding the screening visit (Visit 1);
* Patients who are currently pregnant or planning pregnancy during the study, or lactating;
* Participation in other investigational drug studies or use of other investigational drugs within the previous 30 days prior to randomization;
* History of psychosis;
* A diagnosis of dementia

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2006-05; Primary Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (99):
- United States (32):
  - 248.595.0122 Boehringer Ingelheim Investigational Site, Brimingham, Alabama
  - 248.595.0104 Boehringer Ingelheim Investigational Site, Scottsdale, Arizona
  - 248.595.0133 Boehringer Ingelheim Investigational Site, La Jolla, California
  - 248.595.0140 Boehringer Ingelheim Investigational Site, La Jolla, California
  - 248.595.0112 Boehringer Ingelheim Investigational Site, New Haven, Connecticut
  - 248.595.0113 Boehringer Ingelheim Investigational Site, Bradenton, Florida
  - 248.595.0105 Boehringer Ingelheim Investigational Site, Gainesville, Florida
  - 248.595.0119 Boehringer Ingelheim Investigational Site, Hollywood, Florida
  - 248.595.0124 Boehringer Ingelheim Investigational Site, Palm Beach Gardens, Florida
  - 248.595.0123 Boehringer Ingelheim Investigational Site, Panama City, Florida
  - 248.595.0109 Boehringer Ingelheim Investigational Site, South Miami, Florida
  - 248.595.0115 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 248.595.0106 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 248.595.0103 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 248.595.0127 Boehringer Ingelheim Investigational Site, Augusta, Georgia
  - 248.595.0137 Boehringer Ingelheim Investigational Site, Columbus, Georgia
  - 248.595.0101 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 248.595.0111 Boehringer Ingelheim Investigational Site, Elk Grove Village, Illinois
  - 248.595.0131 Boehringer Ingelheim Investigational Site, Scarbourough, Maine
  - 248.595.0134 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 248.595.0141 Boehringer Ingelheim Investigational Site, Worcester, Massachusetts
  - 248.595.0102 Boehringer Ingelheim Investigational Site, Traverse City, Michigan
  - 248.595.0129 Boehringer Ingelheim Investigational Site, New York, New York
  - 248.595.0139 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 248.595.0136 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 248.595.0120 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 248.595.0107 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 248.595.0118 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 248.595.0114 Boehringer Ingelheim Investigational Site, Warwick, Rhode Island
  - 248.595.0116 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 248.595.0108 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 248.595.0121 Boehringer Ingelheim Investigational Site, Kirkland, Washington
- Austria (5):
  - 248.595.43005 Boehringer Ingelheim Investigational Site, Bruck A. D. Mur
  - 248.595.43003 Boehringer Ingelheim Investigational Site, Graz
  - 248.595.43001 Boehringer Ingelheim Investigational Site, Innsbruck
  - 248.595.43002 Boehringer Ingelheim Investigational Site, Vienna
  - 248.595.43004 Boehringer Ingelheim Investigational Site, Vienna
- Finland (3):
  - 248.595.35803 Boehringer Ingelheim Investigational Site, Helsinki
  - 248.595.35804 Boehringer Ingelheim Investigational Site, Lahti
  - 248.595.35801 Boehringer Ingelheim Investigational Site, Oulu
- France (12):
  - 248.595.3306A Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - 248.595.3306B Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - 248.595.3306C Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - 248.595.3301A Hôpital Gabriel Montpied, Clermont-Ferrand
  - 248.595.3301B Hôpital Gabriel Montpied, Clermont-Ferrand
  - 248.595.3303A Cabinet Médical, Évreux
  - 248.595.3307A Hôpital Roger Salengro, Lille
  - 248.595.3307B Hôpital Roger Salengro, Lille
  - 248.595.3302A Hôpital La Timone, Marseille
  - 248.595.3302B Hôpital La Timone, Marseille
  - 248.595.3305A Hôpital Purpan, Toulouse
  - 248.595.3305C Hôpital Purpan, Toulouse
- Germany (13):
  - 248.595.49006 Boehringer Ingelheim Investigational Site, Augsburg
  - 248.595.49008 Boehringer Ingelheim Investigational Site, Berlin
  - 248.595.49007 Boehringer Ingelheim Investigational Site, Bochum
  - 248.595.49011 Boehringer Ingelheim Investigational Site, Bonn
  - 248.595.49016 Boehringer Ingelheim Investigational Site, Gera
  - 248.595.49009 Boehringer Ingelheim Investigational Site, Göttingen
  - 248.595.49004 Boehringer Ingelheim Investigational Site, Hamburg
  - 248.595.49010 Boehringer Ingelheim Investigational Site, Hanau
  - 248.595.49005 Boehringer Ingelheim Investigational Site, Hanover
  - 248.595.49012 Boehringer Ingelheim Investigational Site, Leipzig
  - 248.595.49001 Boehringer Ingelheim Investigational Site, Marburg
  - 248.595.49015 Boehringer Ingelheim Investigational Site, München
  - 248.595.49014 Boehringer Ingelheim Investigational Site, Tübingen
- Italy (13):
  - 248.595.39004 Università degli Studi di Bari, Bari
  - 248.595.39009 Ospedale di Bellaria, Bologna
  - 248.595.39005 Ospedale della Misericordia, Grosseto
  - 248.595.39001 Azienda Ospedaliera Istituti Clinici di Perfezionamento, Milan
  - 248.595.39010 Ospedale Maggiore Policlinico Mangigalli e Regina Elena, Milan
  - 248.595.39011 Ospedale S. Raffaele - IRCCS, Milan
  - 248.595.39002 Università Federico II, Napoli
  - 248.595.39012 Azienda Ospedaliera Pisana- Università degli Studi di Pisa, Pisa
  - 248.595.39014 Boehringer Ingelheim Investigational Site, Roma
  - 248.595.39006 Policlinico Universitario Molinette, Torino
  - 248.595.39007 Ospedale Evangelico Valdese, Torino
  - 248.595.39013 Ospedale Umberto I, Venezia Mestre
  - 248.595.39003 Ospedale di Viareggio, Viareggio
- Japan (2):
  - 248.595.81001 Juntendo University Hospital, Bunkyo-ku, Tokyo
  - 248.595.81002 Kagawa Prefectural Central Hospital, Takamatsu, Kagawa
- Spain (5):
  - 248.595.34003 Hospital de Alcorcon, Alcorcon (Madrid)
  - 248.595.34001 Hospital Clinic i Provincial of Barcelona, Barcelona
  - 248.595.34002 Nuevo Hospital de Sant Pau, Barcelona
  - 248.595.34004 Hospital 12 de Octubre, Madrid
  - 248.595.34005 Hospital Mutua de Terrassa, Tarrasa (Barcelona)
- Sweden (6):
  - 248.595.46004 Boehringer Ingelheim Investigational Site, Jönköping
  - 248.595.46006 Boehringer Ingelheim Investigational Site, Linköping
  - 248.595.46005 Boehringer Ingelheim Investigational Site, Norrköping
  - 248.595.46002 Boehringer Ingelheim Investigational Site, Örebro
  - 248.595.46001 Boehringer Ingelheim Investigational Site, Stockholm
  - 248.595.46007 Boehringer Ingelheim Investigational Site, Stockholm
- United Kingdom (8):
  - 248.595.44003 Boehringer Ingelheim Investigational Site, Birmingham
  - 248.595.44008 Boehringer Ingelheim Investigational Site, Glasgow
  - 248.595.44004 Boehringer Ingelheim Investigational Site, London
  - 248.595.44002 Boehringer Ingelheim Investigational Site, Newark
  - 248.595.44001 Boehringer Ingelheim Investigational Site, Newcastle upon Tyne
  - 248.595.44010 Boehringer Ingelheim Investigational Site, North Shields
  - 248.595.44011 Boehringer Ingelheim Investigational Site, Romford
  - 248.595.44005 Boehringer Ingelheim Investigational Site, Stoke-on-Trent

REFERENCES:
- [Derived] Schapira AH, McDermott MP, Barone P, Comella CL, Albrecht S, Hsu HH, Massey DH, Mizuno Y, Poewe W, Rascol O, Marek K. Pramipexole in patients with early Parkinson's disease (PROUD): a randomised delayed-start trial. Lancet Neurol. 2013 Aug;12(8):747-55. doi: 10.1016/S1474-4422(13)70117-0. Epub 2013 May 31. PMID 23726851

RESULTS

PARTICIPANT FLOW:
Groups:
- Early Pramipexole: Patients initially randomized to pramipexole were up-titrated from 0.375 mg pramipexole daily to 0.75 mg pramipexole daily and then to 1.5 mg pramipexole daily over a 6 week period, and then 1.5 mg pramipexole daily was continued for the remainder of the 15 months of the study.
- Delayed Pramipexole: Patients initially randomized to placebo, received placebo for 6-9 months, then up-titrated from 0.375 mg pramipexole daily to 1.5 mg pramipexole daily over a 6 week period. These patients were then continued on 1.5 mg pramipexole daily for the remainder of the 15 months of the study.
Period: Overall Study
Arm/Group | Early Pramipexole | Delayed Pramipexole
Started | 261 | 274
Completed | 198 | 192
Not Completed | 63 | 82
Not completed — Adverse Event | 41 | 43
Not completed — Lack of Efficacy | 9 | 14
Not completed — Protocol Violation | 6 | 5
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 6 | 17
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Early Pramipexole: 1.5 milligrams/day pramipexole (for up to 15 months)
- Delayed Pramipexole: Placebo (for first 6 to 9 months) + 1.5 milligrams/day pramipexole (for following 6 months)
- Total: Total of all reporting groups
Arm/Group | Early Pramipexole | Delayed Pramipexole | Total
Number analyzed (Participants) | 261 | 274 | 535
Age, Continuous [Mean (Standard Deviation); unit: Years] — Treated set (TS)
  Years | 62.1 (10.1) | 62.9 (9.9) | 62.5 (10)
Sex: Female, Male [Count of Participants; unit: Participants] — Treated set (TS)
  Participants
    Female | 84 | 108 | 192
    Male | 177 | 166 | 343

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Blinded Rater Unified Parkinson's Disease Rating Scale (UPDRS) Total Score at Month 15
Description: The UPDRS total score (Parts I+II+III) measures the impact of PD on mentation, behaviour and mood, activities of daily living and motor skills on an ordinal scale ranging from 0 (no disability) to 176 (worst disability)
Time Frame: Baseline and Month 15
Population: The Phase 2 Full Analysis Set (FAS2) was made up of all treated participants with a baseline and on-treatment blinded rater assessment of the UPDRS during Phase 2 of the trial
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 211 | 200
Units on a scale | 0.3 (0.7) | 0.7 (0.7)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.6503, ANCOVA; Mean Difference (Net) = -0.4, 95% CI [-2.2 to 1.4], Standard Error of Mean 0.9

2. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Total Score at Month 15
Description: as for outcome 1
Time Frame: Baseline and Month 15
Population: The FAS2 was made up of all treated participants with a baseline and on-treatment blinded rater assessment of the UPDRS during Phase 2 of the trial. 1 patient from the FAS2 was excluded due to insufficient efficacy data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 200
Units on a scale | 0.6 (0.7) | 0.5 (0.7)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.9568, ANCOVA; Mean Difference (Net) = 0.0, 95% CI [-1.7 to 1.8], Standard Error of Mean 0.9

3. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Total Score at Month 9
Description: as for outcome 1
Time Frame: Baseline and Month 9
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 200
Units on a scale | -0.5 (0.6) | 4.3 (0.6)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -4.8, 95% CI [-6.3 to -3.2], Standard Error of Mean 0.8

4. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Total Score at Month 6
Description: as for outcome 1
Time Frame: Baseline and Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 200
Units on a scale | -1.8 (0.6) | 2.6 (0.6)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -4.4, 95% CI [-5.8 to -3], Standard Error of Mean 0.7

5. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Total Score at Month 3
Description: as for outcome 1
Time Frame: Baseline and Month 3
Population: The FAS2 was made up of all treated participants with a baseline and on-treatment blinded rater assessment of the UPDRS during Phase 2 of the trial. 3 patients from the FAS2 were excluded due to insufficient efficacy data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 198
Units on a scale | -2.9 (0.5) | -0.1 (0.5)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -2.9, 95% CI [-4.1 to -1.7], Standard Error of Mean 0.6

6. Secondary Outcome: Change From Baseline in the Blinded Rater UPDRS Parts II+III Total Score at Month 15
Description: The UPDRS Parts II+III total score measures the impact of PD on activities of daily living and motor skills on an ordinal scale ranging from 0 (no disability) to 160 (worst disability)
Time Frame: Baseline and Month 15
Population: The FAS2 was made up of all treated participants with a baseline and on-treatment blinded rater assessment of the UPDRS during Phase 2 of the trial
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 211 | 200
Units on a scale | 0.6 (0.7) | 0.7 (0.7)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.8693, ANCOVA; Mean Difference (Net) = -0.1, 95% CI [-1.8 to 1.5], Standard Error of Mean 0.9

7. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Parts II+III Score at Month 15
Description: as for outcome 6
Time Frame: Baseline and Month 15
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 200
Units on a scale | 0.8 (0.7) | 0.6 (0.7)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.8155, ANCOVA; Mean Difference (Net) = 0.2, 95% CI [-1.5 to 1.9], Standard Error of Mean 0.9

8. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Parts II+III Score at Month 9
Description: as for outcome 6
Time Frame: Baseline and Month 9
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 200
Units on a scale | -0.3 (0.6) | 4.2 (0.6)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -4.5, 95% CI [-6 to -3], Standard Error of Mean 0.8

9. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Parts II+III Score at Month 6
Description: as for outcome 6
Time Frame: Baseline and Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 200
Units on a scale | -1.5 (0.6) | 2.5 (0.6)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -4, 95% CI [-5.4 to -2.6], Standard Error of Mean 0.7

10. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Parts II+III Score at Month 3
Description: as for outcome 6
Time Frame: Baseline and Month 3
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 198
Units on a scale | -2.8 (0.5) | 0.0 (0.5)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -2.8, 95% CI [-3.9 to -1.7], Standard Error of Mean 0.6

11. Secondary Outcome: Change From Baseline in the Blinded Rater UPDRS Part III Total Score at Month 15
Description: The UPDRS Part III total score measures the impact of PD on motor skills on an ordinal scale ranging from 0 (no disability) to 108 (worst disability)
Time Frame: Baseline and Month 15
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 211 | 200
Units on a scale | 0.1 (0.5) | 0.3 (0.5)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.7999, ANCOVA; Mean Difference (Net) = -0.2, 95% CI [-1.5 to 1.1], Standard Error of Mean 0.7

12. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Part III Score at Month 15
Description: as for outcome 11
Time Frame: Baseline and Month 15
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 200
Units on a scale | 0.2 (0.5) | -0.1 (0.5)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.7395, ANCOVA; Mean Difference (Net) = 0.2, 95% CI [-1.1 to 1.5], Standard Error of Mean 0.7

13. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Part III Score at Month 9
Description: as for outcome 11
Time Frame: Baseline and Month 9
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 200
Units on a scale | -0.6 (0.5) | 2.7 (0.5)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -3.3, 95% CI [-4.5 to -2.2], Standard Error of Mean 0.6

14. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Part III Score at Month 6
Description: as for outcome 11
Time Frame: Baseline and Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 200
Units on a scale | -1.6 (0.4) | 1.3 (0.4)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -2.9, 95% CI [-4 to -1.8], Standard Error of Mean 0.6

15. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Part III Score at Month 3
Description: as for outcome 11
Time Frame: Baseline and Month 3
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 198
Units on a scale | -2.1 (0.4) | -0.3 (0.4)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Net) = -1.8, 95% CI [-2.7 to -0.9], Standard Error of Mean 0.5

16. Secondary Outcome: Change From Baseline in the Blinded Rater UPDRS Part II Total Score at Month 15
Description: The UPDRS Part II total score measures the impact of PD on activities of daily living on an ordinal scale ranging from 0 (no disability) to 52 (worst disability)
Time Frame: Baseline and Month 15
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 211 | 200
Units on a scale | 0.5 (0.2) | 0.4 (0.2)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.9256, ANCOVA; Mean Difference (Net) = 0, 95% CI [-0.6 to 0.6], Standard Error of Mean 0.3

17. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Part II Score at Month 15
Description: as for outcome 16
Time Frame: Baseline and Month 15
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 200
Units on a scale | 0.6 (0.2) | 0.6 (0.2)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.9792, ANCOVA; Mean Difference (Net) = 0, 95% CI [-0.6 to 0.6], Standard Error of Mean 0.3

18. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Part II Score at Month 9
Description: as for outcome 16
Time Frame: Baseline and Month 9
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 200
Units on a scale | 0.4 (0.2) | 1.5 (0.2)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Net) = -1.1, 95% CI [-1.7 to -0.5], Standard Error of Mean 0.3

19. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Part II Score at Month 6
Description: as for outcome 16
Time Frame: Baseline and Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 200
Units on a scale | 0.1 (0.2) | 1.2 (0.2)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -1.1, 95% CI [-1.6 to -0.6], Standard Error of Mean 0.3

20. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Part II Score at Month 3
Description: as for outcome 16
Time Frame: Baseline and Month 3
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 198
Units on a scale | -0.7 (0.2) | 0.3 (0.2)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -1, 95% CI [-1.5 to -0.6], Standard Error of Mean 0.2

21. Secondary Outcome: Change From Baseline in the Blinded Rater UPDRS Part I Total Score at Month 15
Description: The UPDRS Part I total score measures the impact of PD on mentation, behaviour and mood on an ordinal scale ranging from 0 (no disability) to 16 (worst disability)
Time Frame: Baseline and Month 15
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 211 | 200
Units on a scale | -0.3 (0.1) | 0 (0.1)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.0376, ANCOVA; Mean Difference (Net) = -0.3, 95% CI [-0.5 to 0], Standard Error of Mean 0.1

22. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Part I Total Score at Month 15
Description: as for outcome 21
Time Frame: Baseline and Month 15
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 200
Units on a scale | -0.2 (0.1) | -0.1 (0.1)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.1607, ANCOVA; Mean Difference (Net) = -0.2, 95% CI [-0.4 to 0.1], Standard Error of Mean 0.1

23. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Part I Total Score at Month 9
Description: as for outcome 21
Time Frame: Baseline and Month 9
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 200
Units on a scale | -0.2 (0.1) | 0.1 (0.1)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.0173, ANCOVA; Mean Difference (Net) = -0.3, 95% CI [-0.5 to -0.1], Standard Error of Mean 0.1

24. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Part I Total Score at Month 6
Description: as for outcome 21
Time Frame: Baseline and Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 200
Units on a scale | -0.3 (0.1) | 0.1 (0.1)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.0007, ANCOVA; Mean Difference (Net) = -0.4, 95% CI [-0.6 to -0.2], Standard Error of Mean 0.1

25. Secondary Outcome: Change From Baseline in the Investigator Rated UPDRS Part I Total Score at Month 3
Description: as for outcome 21
Time Frame: Baseline and Month 3
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 198
Units on a scale | -0.2 (0.1) | -0.1 (0.1)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.4381, ANCOVA; Mean Difference (Net) = -0.1, 95% CI [-0.3 to 0.1], Standard Error of Mean 0.1

26. Secondary Outcome: Number of Responders Using the Blinded Rater Assessment of Clinical Global Impressions of Global Improvement (CGI-I) Score at Month 15
Description: The CGI-I measures the overall improvement in the participants condition from baseline on an ordinal scale ranging from 1 (very much improved) to 7 (very much worse). Responders are defined as those patients with a CGI-I of 1 or 2.
Time Frame: Month 15
Population: The FAS2 was made up of all treated participants with a baseline and on-treatment blinded rater assessment of the UPDRS during Phase 2 of the trial. 27 patients from the FAS2 were excluded due to insufficient CGI-I data.
Measure: Number; unit: Participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 200 | 184
Participants | 18 | 21
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.5116, Regression, Logistic; Odds Ratio (OR) = 0.796, 95% CI [0.403 to 1.573]

27. Secondary Outcome: Change From Baseline in Blinded Rater Assessment of Clinical Global Impressions of Severity of Illness (CGI-S) Category at Month 15
Description: The CGI-S measures the participants severity of illness on an ordinal scale ranging from 1 (normal) to 7 (extremely ill). At Month 15 participants were categorised to 'Improved' (>1 category improvement), 'Unchanged' or 'Worsened' (>1 category worsening).
Time Frame: Baseline and Month 15
Population: The FAS2 was made up of all treated participants with a baseline and on-treatment blinded rater assessment of the UPDRS during Phase 2 of the trial. 4 patients from the FAS2 were excluded due to insufficient CGI-I data.
Measure: Number; unit: Participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 209 | 198
Participants
  Improved | 4 | 3
  Essentially unchanged | 200 | 191
  Worsened | 5 | 4
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; The ordinal responses (3 levels) were analysed using the proportional odds model extension of logistic regression; Test type: Superiority or Other; p = 0.7913, Regression, Logistic; Odds Ratio (OR) = 1.153, 95% CI [0.403 to 3.299]

28. Secondary Outcome: Change From Baseline in the Beck Depression Inventory-Version 1A (BDI-IA) Total Score at Month 15
Description: The BDI measures symptoms of depression on an ordinal scale ranging from 0 (no symptoms) to 63 (worst symptoms)
Time Frame: Baseline and Month 15
Population: The FAS2 was made up of all treated participants with a baseline and on-treatment blinded rater assessment of the UPDRS during Phase 2 of the trial. 3 patients from the FAS2 were excluded due to insufficient BDI data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 211 | 197
Units on a scale | -1 (0.3) | -0.5 (0.3)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.1702, ANCOVA; Mean Difference (Net) = -0.5, 95% CI [-1.3 to 0.2], Standard Error of Mean 0.4

29. Secondary Outcome: Change From Baseline in the Beck Depression Inventory-Version 1A (BDI-IA) Total Score at Month 9
Description: The BDI measures symptoms of depression on an ordinal scale ranging from 0 (no symptoms) to 63 (worst symptoms)
Time Frame: Baseline and Month 9
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 211 | 199
Units on a scale | -1.1 (0.3) | 0.3 (0.3)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.0009, ANCOVA; Mean Difference (Net) = -1.4, 95% CI [-2.2 to -0.6], Standard Error of Mean 0.4

30. Secondary Outcome: Change From Baseline in the Beck Depression Inventory-Version 1A (BDI-IA) Total Score at Month 6
Description: The BDI measures symptoms of depression on an ordinal scale ranging from 0 (no symptoms) to 63 (worst symptoms)
Time Frame: Baseline and Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 211 | 199
Units on a scale | -1.2 (0.3) | 0.2 (0.3)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.0005, ANCOVA; Mean Difference (Net) = -1.4, 95% CI [-2.1 to -0.6], Standard Error of Mean 0.4

31. Secondary Outcome: Change From Baseline in the Beck Depression Inventory-Version 1A (BDI-IA) Total Score at Month 3
Description: The BDI measures symptoms of depression on an ordinal scale ranging from 0 (no symptoms) to 63 (worst symptoms)
Time Frame: Baseline and Month 3
Population: The FAS2 was made up of all treated participants with a baseline and on-treatment blinded rater assessment of the UPDRS during Phase 2 of the trial. 2 patients from the FAS2 were excluded due to insufficient efficacy data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 211 | 198
Units on a scale | -1 (0.3) | -0.3 (0.3)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.0422, ANCOVA; Mean Difference (Net) = -0.7, 95% CI [-1.4 to 0], Standard Error of Mean 0.3

32. Secondary Outcome: Change From Baseline in the Parkinson's Disease Questionnaire-39 (PDQ-39) Overall Index Score at Month 15
Description: The PDQ-39 measures aspects of health in PD participants, the overall index score is the mean of the eight individual domain scores measured on a continuous scale ranging from 0 (no problem at all) to 100 (maximum level of the problem)
Time Frame: Baseline and Month 15
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 211 | 200
Units on a scale | -0.4 (-0.4) [-3.2 to 3.8] | 0.3 (0.3) [-3.6 to 4.4]
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.2149, Wilcoxon (Mann-Whitney); Median Difference (Net) = -0.573, 95% CI [-1.823 to 0.677]

33. Secondary Outcome: Change From Baseline in the Parkinson's Disease Questionnaire-39 (PDQ-39) Overall Index Score at Month 9
Description: as for outcome 32
Time Frame: Baseline and Month 9
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 209 | 199
Units on a scale | -0.5 (-0.5) [-3.6 to 2.0] | 1.4 (1.4) [-2.2 to 5.0]
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.0001, Wilcoxon (Mann-Whitney); Median Difference (Net) = -2.031, 95% CI [-3.125 to -0.938]

34. Secondary Outcome: Change From Baseline in the European Quality of Life Scale (EUROQOL (EQ)-5D) Overall Index Score at Month 15
Description: The EQ-5D measures health status on a continuous scale ranging from 0 (dead) to 1 (full health)
Time Frame: Baseline and Month 15
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 200
Units on a scale | 0 (0) [-0.026 to 0.092] | 0 (0) [-0.079 to 0.078]
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.2605, Wilcoxon (Mann-Whitney); Median Difference (Net) = 0, 95% CI [0 to 0.026]

35. Secondary Outcome: Change From Baseline in the European Quality of Life Scale (EUROQOL (EQ)-5D) Overall Index Score at Month 9
Description: The EQ-5D measures health status on a continuous scale ranging from 0 (dead) to 1 (full health)
Time Frame: Baseline and Month 9
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 209 | 199
Units on a scale | 0 (0) [-0.026 to 0.092] | 0 (0) [-0.140 to 0]
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); Median Difference (Net) = 0.051, 95% CI [0 to 0.089]

36. Secondary Outcome: Change From Baseline in the European Quality of Life Visual Analogue Scale (EUROQOL (EQ) VAS) Score at Month 15
Description: The EQ-VAS is a self rating of current health-related quality of life measured on a continuous scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state)
Time Frame: Baseline and Month 15
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 210 | 199
Units on a scale | 0 (0) [-8.0 to 7.0] | 0 (0) [-10.0 to 2.0]
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.0489, Wilcoxon (Mann-Whitney); Median Difference (Net) = 2, 95% CI [0 to 5]

37. Secondary Outcome: Change From Baseline in the European Quality of Life Visual Analogue Scale (EUROQOL (EQ) VAS) Score at Month 9
Description: as for outcome 36
Time Frame: Baseline and Month 9
Population: The FAS2 was made up of all treated participants with a baseline and on-treatment blinded rater assessment of the UPDRS during Phase 2 of the trial. 5 patients from the FAS2 were excluded due to insufficient efficacy data.
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 208 | 198
Units on a scale | 0 (0) [-5.5 to 5.0] | -0.5 (-0.5) [-10.0 to 5.0]
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.0282, Wilcoxon (Mann-Whitney); Median Difference (Net) = 3, 95% CI [0 to 5]

38. Secondary Outcome: Modified Minnesota Disorders Interview (MMIDI) Risk of Gambling at Month 1
Description: The MMIDI is a semi-structured interview designed to assess impulse control disorders; risk of gambling is assessed via 12 questions, a participant is considered at risk if answering 'Yes' to Q1 and 'Yes' to 5 or more of Q2 to Q12.
Time Frame: Month 1
Population: The FAS2 was made up of all treated participants with a baseline and on-treatment blinded rater assessment of the UPDRS during Phase 2 of the trial. 132 patients from the FAS2 were excluded due to insufficient MMIDI data.
Measure: Number; unit: Participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 146 | 133
Participants
  No risk of gambling | 146 | 133
  Risk of gambling | 0 | 0

39. Secondary Outcome: Modified Minnesota Disorders Interview (MMIDI) Risk of Gambling at Month 6
Description: as for outcome 38
Time Frame: Month 6
Population: The FAS2 was made up of all treated participants with a baseline and on-treatment blinded rater assessment of the UPDRS during Phase 2 of the trial. 131 patients from the FAS2 were excluded due to insufficient MMIDI data.
Measure: Number; unit: Participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 146 | 134
Participants
  No risk of gambling | 146 | 134
  Risk of gambling | 0 | 0

40. Secondary Outcome: Modified Minnesota Disorders Interview (MMIDI) Risk of Gambling at Month 9
Description: as for outcome 38
Time Frame: Month 9
Population: as for outcome 39
Measure: Number; unit: Participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 146 | 134
Participants
  No risk of gambling | 146 | 134
  Risk of gambling | 0 | 0

41. Secondary Outcome: Modified Minnesota Disorders Interview (MMIDI) Risk of Gambling at Month 12
Description: as for outcome 38
Time Frame: Month 12
Population: The FAS2 was made up of all treated participants with a baseline and on-treatment blinded rater assessment of the UPDRS during Phase 2 of the trial. 140 patients from the FAS2 were excluded due to insufficient MMIDI data.
Measure: Number; unit: Participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 143 | 128
Participants
  No risk of gambling | 143 | 128
  Risk of gambling | 0 | 0

42. Secondary Outcome: Modified Minnesota Disorders Interview (MMIDI) Risk of Gambling at Month 15
Description: as for outcome 38
Time Frame: Month 15
Population: The FAS2 was made up of all treated participants with a baseline and on-treatment blinded rater assessment of the UPDRS during Phase 2 of the trial. 134 patients from the FAS2 were excluded due to insufficient MMIDI data.
Measure: Number; unit: Participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 145 | 132
Participants
  No risk of gambling | 145 | 132
  Risk of gambling | 0 | 0

43. Secondary Outcome: Modified Minnesota Disorders Interview (MMIDI) for Compulsive Sexual Behaviour at Month 1
Description: The MMIDI is a semi-structured interview designed to assess impulse control disorders; compulsive sexual behaviour is assessed via 4 questions, a participant is considered as being compulsive if answering 'Yes' to Q1 and 'Yes' to 1 or more of Q2 to Q4.
Time Frame: Month 1
Population: as for outcome 38
Measure: Number; unit: Participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 146 | 133
Participants
  No compulsive sexual behaviour | 146 | 133
  Compulsive sexual behaviour | 0 | 0

44. Secondary Outcome: Modified Minnesota Disorders Interview (MMIDI) for Compulsive Sexual Behaviour at Month 6
Description: as for outcome 43
Time Frame: Month 6
Population: as for outcome 39
Measure: Number; unit: Participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 146 | 134
Participants
  No compulsive sexual behaviour | 146 | 134
  Compulsive sexual behaviour | 0 | 0

45. Secondary Outcome: Modified Minnesota Disorders Interview (MMIDI) for Compulsive Sexual Behaviour at Month 9
Description: as for outcome 43
Time Frame: Month 9
Population: as for outcome 39
Measure: Number; unit: Participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 146 | 134
Participants
  No compulsive sexual behaviour | 146 | 134
  Compulsive sexual behaviour | 0 | 0

46. Secondary Outcome: Modified Minnesota Disorders Interview (MMIDI) for Compulsive Sexual Behaviour at Month 12
Description: as for outcome 43
Time Frame: Month 12
Population: as for outcome 41
Measure: Number; unit: Participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 143 | 128
Participants
  No compulsive sexual behaviour | 143 | 126
  Compulsive sexual behaviour | 0 | 2

47. Secondary Outcome: Modified Minnesota Disorders Interview (MMIDI) for Compulsive Sexual Behaviour at Month 15
Description: as for outcome 43
Time Frame: Month 15
Population: as for outcome 42
Measure: Number; unit: Participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 145 | 132
Participants
  No compulsive sexual behaviour | 145 | 131
  Compulsive sexual behaviour | 0 | 1

48. Secondary Outcome: Modified Minnesota Disorders Interview (MMIDI) for Compulsive Buying at Month 1
Description: The MMIDI is a semi-structured interview designed to assess impulse control disorders; compulsive buying is assessed via 4 questions, a participant is considered as being compulsive if answering 'Yes' to Q1a and 'Yes' to 1 or more of Q2a, Q3a and Q4a.
Time Frame: Month 1
Population: as for outcome 38
Measure: Number; unit: Participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 146 | 133
Participants
  No compulsive buying | 145 | 133
  Compulsive buying | 1 | 0

49. Secondary Outcome: Modified Minnesota Disorders Interview (MMIDI) for Compulsive Buying at Month 6
Description: as for outcome 48
Time Frame: Month 6
Population: as for outcome 39
Measure: Number; unit: Participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 146 | 134
Participants
  No compulsive buying | 144 | 134
  Compulsive buying | 2 | 0

50. Secondary Outcome: Modified Minnesota Disorders Interview (MMIDI) for Compulsive Buying at Month 9
Description: as for outcome 48
Time Frame: Month 9
Population: as for outcome 39
Measure: Number; unit: Participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 146 | 134
Participants
  No compulsive buying | 143 | 134
  Compulsive buying | 3 | 0

51. Secondary Outcome: Modified Minnesota Disorders Interview (MMIDI) for Compulsive Buying at Month 12
Description: as for outcome 48
Time Frame: Month 12
Population: as for outcome 41
Measure: Number; unit: Participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 143 | 128
Participants
  No compulsive buying | 141 | 128
  Compulsive buying | 2 | 0

52. Secondary Outcome: Modified Minnesota Disorders Interview (MMIDI) for Compulsive Buying at Month 15
Description: as for outcome 48
Time Frame: Month 15
Population: as for outcome 42
Measure: Number; unit: Participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 145 | 132
Participants
  No compulsive buying | 143 | 132
  Compulsive buying | 2 | 0

53. Secondary Outcome: Percentage Change From Baseline in the Striatum Uptake at Month 15
Description: The striatum beta-carbomethoxy-iodophenyl-tropane (beta-CIT) uptake was calculated as mean of the left and right caudate and putamen regions; measured by the Single-Photon Emission Computed Tomography (SPECT).
Time Frame: Baseline and Month 15
Population: The substudy set was made up of all randomised patients with a baseline and end of treatment assessment of striatal uptake.
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 62 | 61
Percentage change | -15.1 (2.1) | -14.6 (2)
Statistical Analysis 1: Comparison: Early Pramipexole vs Delayed Pramipexole; Test type: Superiority or Other; p = 0.8397, ANCOVA; Mean Difference (Net) = -0.5, 95% CI [-5.4 to 4.4], Standard Error of Mean 2.5

54. Secondary Outcome: Clinically Significant Abnormalities in Clinical Laboratory Measurements - Haematology and Electrolytes
Time Frame: Baseline and Month 15
Population: Treated set: Haematocrit and mean corpuscular volume (MCV-N) was 211 for Early PPX and 209 for Delayed PPX, Haemoglobin-N was 213 for Early PPX and 212 for Delayed PPX, Sodium-N was 211 for Early PPX and 209 for Delayed PPX, Calcium and Chloride-N was 214 for Early PPX and 209 for Delayed PPX, Phosphate-N was 201 for Early and Delayed PPX
Measure: Number; unit: percentage of participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 211 | 209
percentage of participants
  Haematocrit - decrease | 1.4 | 1.0
  Haemoglobin - decrease | 2.3 | 0.9
  MCV - increase | 0.5 | 0
  Sodium - decrease | 1.4 | 0.5
  Calcium - increase | 0 | 0.5
  Chloride - decrease | 0.9 | 0
  Phosphate - decrease | 1.0 | 0
  Phosphate - increase | 0.5 | 0

55. Secondary Outcome: Clinically Significant Abnormalities in Clinical Laboratory Measurements - Enzymes
Time Frame: Baseline and Month 15
Population: Gamma Glutamyltranspeptidase (GGT-N) was 214 for Early PPX and 208 for Delayed PPX, Amylase-N was 214 for Early PPX and 209 for Delayed PPX
Measure: Number; unit: percentage of participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 214 | 209
percentage of participants
  GGT - increase | 0.5 | 0
  Amylase - increase | 1.4 | 0

56. Secondary Outcome: Clinically Significant Abnormalities in Clinical Laboratory Measurements - Substrates
Time Frame: Baseline and Month 15
Population: Glucose-N was 28 for Early PPX and 46 for Delayed PPX, Cholesterol and Triglyceride-N was 213 for Early PPX and 208 for Delayed PPX, Blood Urea Nitrogen-N was 214 for Early PPX and 209 for Delayed PPX, Creatinine-N was 200 for Early PPX and 202 for Delayed PPX, Uric Acid-N was 212 for Early PPX and 209 for Delayed PPX.
Measure: Number; unit: percentage of participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 214 | 209
percentage of participants
  Glucose - decrease | 0 | 2.2
  Glucose - increase | 3.6 | 0
  Cholesterol - increase | 1.4 | 2.9
  Blood Urea Nitrogen - increase | 0.9 | 0.5
  Creatinine - increase | 0.5 | 1.0
  Triglyceride - increase | 1.4 | 0
  Uric acid - increase | 0.5 | 0.5

57. Secondary Outcome: Clinically Significant Abnormalities in Vital Signs
Time Frame: Baseline and Month 15
Population: Phase 1 Treated set for sinus bradycardia with N of 261 for Early PPX and 274 for Delayed PPX. Phase 2 Treated set for hypotension with N of 221 for Early PPX and 214 for Delayed PPX.
Measure: Number; unit: percentage of participants
Arm/Group | Early Pramipexole | Delayed Pramipexole
Number analyzed (Participants) | 261 | 274
percentage of participants
  Sinus bradycardia | 0 | 0.4
  Hypotension | 0 | 0.5

ADVERSE EVENTS:
Time Frame: Onset date after the date of first dose up to 48 hours after last dose of study drug.
Arm/Group | Early Pramipexole | Delayed Pramipexole
Serious Adverse Events (participants affected / at risk) | 25/261 | 25/274
Other Adverse Events (participants affected / at risk) | 172/261 | 164/274
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Pramipexole (N=261) | Delayed Pramipexole (N=274)
Urinary tract infection (Infections and infestations) | 0 | 2
Bacterial infection (Infections and infestations) | 1 | 0
Gastroenteristis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Large cell carcinoma of the respiratory tract stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Pakinson's disease (Nervous system disorders) | 1 | 1
Pakinsonism (Nervous system disorders) | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Macular hole (Eye disorders) | 1 | 0
Pterygium (Eye disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral arterial occulsive disease (Vascular disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Small intestine obstruction (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Breast disorder (Reproductive system and breast disorders) | 1 | 0
Varicocele (Reproductive system and breast disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Hyperplasia (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Radial nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Early Pramipexole (N=261) | Delayed Pramipexole (N=274)
Nasopharyngitis (Infections and infestations) | 19 | 24
Insomnia (Psychiatric disorders) | 26 | 21
Depression (Psychiatric disorders) | 18 | 16
Sleep disorder (Psychiatric disorders) | 14 | 6
Abnormal dreams (Psychiatric disorders) | 8 | 14
Somnolence (Nervous system disorders) | 36 | 21
Dizziness (Nervous system disorders) | 35 | 33
Headache (Nervous system disorders) | 20 | 28
Hypertension (Vascular disorders) | 11 | 16
Nausea (Gastrointestinal disorders) | 62 | 49
Constipation (Gastrointestinal disorders) | 19 | 28
Diarrhoea (Gastrointestinal disorders) | 10 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 6
Fatigue (General disorders) | 36 | 38
Oedema peripheral (General disorders) | 25 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.